CLINICAL TRIAL: NCT00421512
Title: A Phase I Study of Bevacizumab and Sunitinib in Metastatic Renal Cell Carcinoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Robert Motzer, MD, Memorial Sloan Kettering Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-016
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal cell carcinoma; Metastatic; Kidney Cancer; Bevacizumab; Sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Sunitinib

INTERVENTIONS:
Drug: Bevacizumab and Sunitinib — On Cycle 1, Day 0, patients will begin treatment with bevacizumab. Sunitinib will begin on Day 1. The starting dose for sunitinib will be 25mg orally daily. sunitinib will be given in a four weeks on-two weeks off schedule. Bevacizumab will begin on Day 0 and will be administered every two weeks at 10mg/kg. A cycle of therapy is 6 weeks. The sunitinib dose escalation portion of the trial will be performed to determine the MTD of sunitinib given in combination with bevacizumab. Once the MTD has been determined, 10 additional patients will be treated at the MTD of sunitinib in combination with bevacizumab.

SUMMARY:
The purpose of this study is to test the safety of bevacizumab and sunitinib given in combination for kidney cancer. The drugs act to stop blood vessel growth but in different ways. They have not been studied together in a previous study. We also want to find out what effects (good and bad) the combination of bevacizumab and sunitinib have on you and your tumor.

DETAILED DESCRIPTION:
To assess the maximum tolerated dose and overall safety and tolerability of sunitinib administered in combination with bevacizumab for the treatment of patients with metastatic renal cell carcinoma.

To assess antitumor activity of the combination of sunitinib and bevacizumab. To evaluate serum levels of vascular endothelial growth factor (VEGF) in patients treated with sunitinib and bevacizumab.

Study Design: This is a single center, open-label, Phase 1 study of sunitinib in combination with bevacizumab in patients with advanced metastatic renal cell carcinoma. This study is designed to confirm that the two agents can be administered safely in combination. Patients will begin treatment with bevacizumab on Day 0 and sunitinib on Day 1. Bevacizumab will be administered intravenously every two weeks. Sunitinib will be given orally on a 4 weeks on, 2 weeks off schedule. DLT determination will be based on toxicities observed in Cycles 1 - a cycle is defined by sunitinib dosing (6 weeks). Once the MTD for the combination has been identified, 10 additional patients will be enrolled at the MTD to further assess safety and efficacy. Patients will be treated with bevacizumab and sunitinib until there is disease progression, significant toxicity or withdrawal of patient consent. The maximum treatment duration is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma (of any histological subtype) and with metastases. Patients with unresected primary tumors may be enrolled as long as evidence of metastatic disease is also present.
* Evidence of unidimensionally measurable disease (i.e., greater than or equal to 1 malignant tumor mass that can be accurately measured in at least 1 dimension greater than or equal to 20 mm with conventional computerized tomography [CT] or magnetic resonance imaging [MRI], or greater than or equal to 10 mm with spiral CT scan [if spiral CT scan is used, minimum lesion size should be twice the reconstruction interval used, e.g., if reconstruction size is 7 mm, lesion size should be greater than or equal to 14 mm]).
* Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable.
* Male or female, 18 years of age or older.
* ECOG performance status 0 or 1.
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedure to NCI CTCAE grade less than or equal to 1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 1.5 x upper limit of normal (ULN)
* Total serum bilirubin less than or equal to 1.5 mg/dL
* Total white blood cell count greater than or equal to 3000 cells/µL
* Absolute neutrophil count (ANC) greater than or equal to 1500/µL
* Platelets greater than or equal to 100,000/µL
* Hemoglobin greater than or equal to 9.0 g/dL
* Serum calcium less than or equal to 12.0 mg/dL
* Serum creatinine less than or equal to 2.0 x ULN
* PT less than or equal to 1.5 ULN
* Urine protein:creatinine ratio less than or equal to 1.0 at screening
* Negative pregnancy test (only in women of childbearing age)
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Patients eligible for the higher priority IRB protocol #07-066
* Major surgery, open biopsy, traumatic injury, radiation or systemic therapy within 4 weeks of starting the study treatment. Anticipation of major surgical procedure during the study. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* More than 2 prior systemic therapies for metastatic RCC.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* NCI CTCAE grade 3 hemorrhage within the past 1 month.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* History of or known brain metastases, current spinal cord compression, or carcinomatous meningitis.
* Any of the following within the 12 months prior to study drug administration:

  * severe/unstable angina, MI, CABG, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack or peripheral vascular disease.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater than or equal to 2, atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec for males and >470 msec for females.
* Blood pressure > 150/90mmHg
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer or bone fracture
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Current treatment on another therapeutic clinical trial.
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the 7 days prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Receipt of any investigational agent within 4 weeks prior to study entry.
* History of severe hypersensitivity reaction to bevacizumab or to any other component of bevacizumab.
* Prior treatment with sunitinib, bevacizumab
* Prior sorafenib given less than 8 weeks prior to study entry.
* Unresolved symptoms or signs related to sorafenib within 8 weeks prior to study entry.
* Use of therapeutic doses of coumadin.
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose and overall safety and tolerability of sunitinib administered in combination with bevacizumab for the treatment of patients with metastatic renal cell carcinoma. | DLT determination will be based on toxicities observed in Cycles 1

SECONDARY OUTCOMES:
To assess antitumor activity of the combination of sunitinib and bevacizumab. | 28 days +/- 3
To evaluate serum levels of vascular endothelial growth factor (VEGF) | every 28 days of a cycle +/- 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org